CLINICAL TRIAL: NCT06747962
Title: A1 Pulley Release and Pull-out Tenolysis Versus Simple A1 Pulley Release in Trigger Fingers and Thumb. a Randomized Controlled Trial
Brief Title: Pull-out Tenolysis Versus Simple A1 Pulley Release in Trigger Digits
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eleni Karagergou (Other)
Responsible Party: Sponsor-Investigator, Eleni Karagergou, Consultant Plastic and Hand Surgeon, Aristotle University Of Thessaloniki
Organization: Aristotle University Of Thessaloniki (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1543/ 18.11.2024
Record Dates: First submitted 2024-12-19; First posted 2024-12-24 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Trigger Digit
Keywords: trigger finger; trigger thumb; traction tenolysis; pull-out tenolysis; A1 pulley
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pull out tenolysis group (Active Comparator): A1 pulley release and pull out tenolysis for the treatment of trigger fingers and thumb
  Interventions: Procedure: A1 pulley release and pull out tenolysis
- Simple A1 pulley release group (Placebo Comparator): Simple A1 pulley release for the treatment of trigger fingers and thumb
  Interventions: Procedure: Simple A1 pulley release

INTERVENTIONS:
Procedure: A1 pulley release and pull out tenolysis — A short transverse incision will be made over the proximal or distal palmar crease, according to the digit involved. Blunt dissection will be used to spread the subcutaneous tissue and the palmar fascia to expose the A1 pulley. The digital nerves and vessels will be retracted and protected. The proximal edge of the A1 pulley will be identified and a scalpel blade will be used to divide the entire A1 pulley under direct vision. Flexor digitorum superficialis and flexor digitorum profundus tendons or flexor pollicis longus tendon (for the thumb) will be gently pulled out of the wound with two mosquito forceps to break any adhesions. The wound will be closed primarily with sutures. The patient will be asked to actively move the digit to confirm complete relief of triggering.The wound will be closed primarily with sutures.
  Arms: Pull out tenolysis group
Procedure: Simple A1 pulley release — A short transverse incision will be made over the proximal or distal palmar crease, according to the digit involved. Blunt dissection will be used to spread the subcutaneous tissue and the palmar fascia to expose the A1 pulley. The digital nerves and vessels will be retracted and protected. The proximal edge of the A1 pulley will be identified and a scalpel blade will be used to divide the entire A1 pulley vision. After release, the patient will be asked to actively move the digit to confirm complete relief of triggering.The wound will be closed primarily with sutures.
  Arms: Simple A1 pulley release group

SUMMARY:
Trigger finger is a common tendinopathy and clinically presents with painful catching or popping as the patient flexes and extends the digit, due to mechanical impingement of the thickened flexor tendons as they pass through a narrow tendon sheath canal at the level of the metacarpal head. If conservative management with corticosteroid injection and splinting fails or if symptoms recur, surgery and division of the A1 pulley are indicated. Traction (or pull- out) tenolysis is a maneuver based on pulling of the flexor tendons out of the wound, to release any adhesions that might have occurred due to long- standing triggering. Although it has been associated with postoperative pain and stiffness, no robust evidence exists to support its benefit or not. In view of the low quality evidence regarding the pros and cons of traction (or pull-out) tenolysis following A1 pulley release, the investigators will compare simple A1 pulley release versus A1 pulley release and pull-out tenolysis in a prospective randomized study design. Hypothesis of the study is that the pull- out tenolysis yields better results in terms of total active range of movement, pinch and grip strength, pain and quick-DASH scoring when compared to simple pulley release. The confirmation of the hypothesis will justify the use of pull-out tenolysis as a means of breaking any tendon adhesions and returning to normal function sooner. On the contrary, if the pull-out tenolysis is linked to a less favorable functional outcome, simple A1 pulley release will be recommended.

DETAILED DESCRIPTION:
Trigger finger is a common condition that can cause hand pain and disability. It involves entrapment of the flexor tendons of the fingers and thumb within their flexor tendon sheath at the level of the metacarpal head. This phenomenon is due to the mechanical impingement of the thickened flexor tendons as they pass through a narrow tendon sheath canal. It can cause painful catching or popping as the patient flexes and extends the digit. On occasion, the digit will lock in flexion and require passive manipulation to extend. Initial management can be conservative with corticosteroid injection and splinting. If conservative management fails or if symptoms recur, surgical release of the A1 pulley is indicated. This is a common procedure which is performed under local anaesthesia. Intraoperatively, following division of A1 pulley, a traction tenolysis is occasionally performed by some surgeons. This maneuver, which is based on pulling of the flexor tendons out of the wound, is believed to release any adhesions that might have occurred due to long- standing triggering but it has been reported to result in prolonged postoperative pain and stiffness. However, there is no robust evidence to support a less favorable outcome following traction tenolysis. Aim of the study: In view of the low quality evidence regarding the pros and cons of traction (or pull-out) tenolysis following A1 pulley release, the investigators will compare simple A1 pulley release versus A1 pulley release and pull-out tenolysis in a prospective randomized study design. Hypothesis of the study is that the pull-out tenolysis yields better results in terms of total active range of movement, pinch and grip strength, pain and quick-DASH scoring when compared to simple pulley release. The confirmation of the hypothesis will justify the use of pull-out tenolysis as a means of breaking any tendon adhesions and returning to normal function sooner. On the contrary, if the pull- out tenolysis is linked to a less favorable functional outcome, simple A1 pulley release will be recommended. The study will be conducted in accordance with the Declaration of Helsinki and the Guidelines on Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with single trigger finger that failed conservative treatment
* Patients with single trigger finger that had recurrence of symptoms after conservative treatment

Exclusion Criteria:

* Patients with limited range of movement before appearance of triggering
* Patients with osteoarthritis / rheumatoid arthritis
* Patients that had a second procedure at the same time of trigger finger release (eg carpal tunnel release).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Total active range of motion (AROM) of the affected finger | 2 weeks
  Comparison of total (AROM) between the groups. Measurements will be done with a goniometer
Total active range of motion (AROM) of the affected finger | 6 weeks
  Comparison of total (AROM) between the groups. Measurements will be done with a goniometer.
Total active range of motion (AROM) of the affected finger | 3 months
  Comparison of total (AROM) between the groups. Measurements will be done with a goniometer.
Visual Analog Scale (VAS) for pain relief | 2 weeks
  Comparison of the VAS for pain between the groups. Minimum 0, Maximum 10, higher scores mean a worse outcome
Visual Analog Scale (VAS) for pain relief | 6 weeks
  Comparison of the VAS for pain between the groups. Minimum 0, Maximum 10, higher scores mean a worse outcome
Visual Analog Scale (VAS) for pain relief | 3 months
  Comparison of the VAS for pain between the groups. Minimum 0, Maximum 10, higher scores mean a worse outcome

SECONDARY OUTCOMES:
Grip and Pinch strength | 6 weeks
  Comparison of grip and pinch strength between the groups, as measured by a dynamometer
Grip and Pinch strength | 3 months
  Comparison of grip and pinch strength between the groups, as measured by a dynamometer
Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) functional score | 6 weeks
  Comparison of the QuickDASH score between the two groups. Minimum 0, Maximum 100, higher scores mean a worse outcome.
Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) functional score | 3 months
  Comparison of the QuickDASH score between the two groups. Minimum 0, Maximum 100, higher scores mean a worse outcome.

OTHER OUTCOMES:
Rate of complications | Up to 3 months postoperatively
  All complications, such as swelling, wound dehiscence and infection, will be documented and rates will be compared between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Givissis, Professor, Study Chair — Aristotle University Of Thessaloniki
Locations (1):
- Aristotle University of Thessaloniki, 1st Orthopaedic Department, G. Papanikolaou Hospital, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choudhury MM, Tay SC. Outcome of traction tenolysis in open trigger finger release--a retrospective review. Hand Surg. 2013;18(3):375-9. doi: 10.1142/S0218810413500421. PMID 24156581
- [Background] Baek JH, Chung DW, Lee JH. Factors Causing Prolonged Postoperative Symptoms Despite Absence of Complications After A1 Pulley Release for Trigger Finger. J Hand Surg Am. 2019 Apr;44(4):338.e1-338.e6. doi: 10.1016/j.jhsa.2018.06.023. Epub 2018 Jul 25. PMID 30054030
- [Background] Yang TC, Fufa D, Huang HK, Huang YC, Chang MC, Wang JP. Percutaneous A1 Pulley Release Combined with Finger Splint for Trigger Finger with Proximal Interphalangeal Joint Flexion Contracture. J Hand Surg Asian Pac Vol. 2019 Sep;24(3):270-275. doi: 10.1142/S2424835519500334. PMID 31438789